CLINICAL TRIAL: NCT00984178
Title: Randomized Trial Comparing Intracoronary Delivery of Bone Marrow-derived Stem Cells Versus Stem Cell Mobilisation With GCSF, a Combination of Both Therapies and Conventional Treatment in Patients With Reperfused Acute Myocardial Infarction
Brief Title: Trial of Hematopoietic Stem Cells in Acute Myocardial Infarction
Acronym: TECAM2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TECAM Group (Network)
Collaborators: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Francisco Fernández-Avilés, TECAM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-005149-36; PI041078
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-09

CONDITIONS: Reperfused Acute Myocardial Infarction
Keywords: Reperfusion; acute myocardial infarction; stem cell therapy; GCSF; bone marrow mononuclear cells; magnetic resonance
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention): standard treatment
- Bone marrow mononuclear progenitors (Experimental): intracoronary transplantation of bone-marrow mononuclear progenitor cells
  Interventions: Other: Bone marrow mononuclear cells
- GCSF (Experimental): progenitor cells mobilization through Granulocite- Colony Stimulating Factor treatment (G-CSF)
  Interventions: Other: Granulocite Colony Stimulating Factor treatment (G-CSF)
- GCSF plus bone marrow mononuclear cells (Experimental): combined treatment (intracoronary transplantation plus cell mobilization with G-CSF).
  Interventions: Other: Granulocite Colony Stimulating Factor treatment (G-CSF); Other: Bone marrow mononuclear cells

INTERVENTIONS:
Other: Granulocite Colony Stimulating Factor treatment (G-CSF) — G-CSF will be administered at a dose of 10 mcg/kg/day. The administration begins at the first 24 hours post-reperfusion, remaining for 5 days
  Arms: GCSF; GCSF plus bone marrow mononuclear cells
Other: Bone marrow mononuclear cells — Bone marrow mononuclear cells will be isolated with a Ficoll technique from 50 cc of bone marrow aspiration
  Arms: Bone marrow mononuclear progenitors; GCSF plus bone marrow mononuclear cells

SUMMARY:
The aim of this study is to compare the effectiveness of four different strategies for preventing the ventricular postinfarction remodelling: 1) Conventional treatment for reperfunded extensive acute myocardial infarction, 2) Autologous bone marrow stem-cells intracoronary transplantation 3) mobilization of bone marrow stem-cells induced by granulocyte colony-stimulating factors (G-CSF); and 4) combined treatment (stem-cells transplantation plus mobilization with G-CSF).

DETAILED DESCRIPTION:
This clinical study is a phase II randomized trial for patients with an acute extensive reperfunded myocardial infarction who undergo coronary artery revascularization with sirolimus coated stents. The aim of this study is to compare the effectiveness of four different strategies for preventing the ventricular postinfarction remodelling: 1) Conventional treatment for reperfunded extensive acute myocardial infarction, 2) Autologous bone marrow stem-cells intracoronary transplantation 3) mobilization of bone marrow stem-cells induced by granulocyte colony-stimulating factors (G-CSF); and 4) combined treatment (stem-cells transplantation plus mobilization with G-CSF). The investigational follow-up will be at 30 days, 4 and 9 months.Effectiveness of the therapies on neomyogenesis will be measured by Magnetic Resonance Imaging analysis of left ventricular size and global and regional function and the myocardial viability.The impact of the therapies on stent re-endothelialization and restenosis will be analysed by angiography and intracoronary ultrasounds at 30 days and 9 months. The impact of the different treatments on neoangiogenesis will be measured by infarct related artery intracoronary study of the evolution of coronary flow reserve. Also, it will be measured the haematopoietic precursors kinetic in the different treatment branches.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Acute myocardial infarction with the following characteristics:

  * Clinical symptoms of chest pain lasting >30 minutes, unresponsive to nitroglycerin.
  * Typical myocardial enzymatical necrotic curve
  * Total summed ST-segment elevation ≥ 6 mm in 12-lead electrocardiogram.
* Akynesis or hypokinesis in infarct-related artery area without contractility abnormalities in the rest of areas.
* Pharmacological, mechanical or both type reperfusions (facilitated angioplasty) with evidence of normal infarcted area epicardial flow (TIMI grade 3) in the first 24 hours after the beginning of the symptoms
* Successful repair of the infarct-related artery (residual post-stenting stenosis < 30% by visual estimation with epicardial normal flow [grade 3] in the first 24 hours after the beginning of the symptoms or lack of significant residual lesions evidence (<50% visual estimation) in infarct-related artery.
* Lack of evidence of significant lesions in the remaining coronary vessels or adequate revascularization achieved in the first 24 hours after symptoms began.

Exclusion Criteria:

* The presence of cardiogenic shock defined as sustained systolic blood pressure less than 90 mm Hg, with no response to fluids or systolic blood pressure less than 100 mm Hg with vasopressors (in absence of bradycardia)
* Suspicion or evidence of infarct mechanical complication
* History of sustained ventricular tachycardia or atrial fibrillation
* Patient with cardiac defibrillator or candidate for its potential implantation.
* Investigational drug treatment in the previous 4 weeks
* Actual or potential use of anti-neoplastic drugs
* Oncology antecedents in the last 5 years
* Previous treatment with trans myocardial laser revascularization
* Women of childbearing potential
* Severe concomitant disease modifying patient's survival during the study
* Inability to suspend thrombolytic treatment
* Active bleeding or major surgery within 2 weeks forbidding the use of heparin, abciximab or antiplatelet therapy.
* Previous malignant haematology disease (leukaemia or lymphomas) or hypercoagulability disorders (antiphospholipid syndrome, antithrombin, C-protein and S-protein or V Leiden Factor deficiency)
* Previous known renal failure (creatinine > 2.5 mg /dl)
* Any kind of stroke in the last year or whenever episode of haemorrhagic stroke.
* Major surgery pending in the next year
* Previously known vascular disease that prevents from catheterization.
* Evidence of hypersensitivity to Filgrastim, proteins derived from E. coli or any formulation component.
* Inability to give written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
The change in left ventricular ejection fraction and left ventricular end-systolic volume relative to baseline measured by magnetic resonance | 9 months

SECONDARY OUTCOMES:
The change in left ventricle end-dyastolyc volume, segment contractility, wall thickness and intravascular ultrasound reendothelization relative to baseline measured by magnetic resonance and other imaging techniques | 9 months
To determine the safety of the study procedures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernandez-Aviles, MD, PhD, Study Chair — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital Universitario de Valladolid, Valladolid, Valladolid, Spain

REFERENCES:
- [Derived] San Roman JA, Sanchez PL, Villa A, Sanz-Ruiz R, Fernandez-Santos ME, Gimeno F, Ramos B, Arnold R, Serrador A, Gutierrez H, Martin-Herrero F, Rollan MJ, Fernandez-Vazquez F, Lopez-Messa J, Ancillo P, Perez-Ojeda G, Fernandez-Aviles F. Comparison of Different Bone Marrow-Derived Stem Cell Approaches in Reperfused STEMI. A Multicenter, Prospective, Randomized, Open-Labeled TECAM Trial. J Am Coll Cardiol. 2015 Jun 9;65(22):2372-82. doi: 10.1016/j.jacc.2015.03.563. PMID 26046730
- See also: Webmail of the TECAM group — http://www.cardiovascularcelltherapy.com/